CLINICAL TRIAL: NCT04664595
Title: Requirements of Propofol With Target Controlled Infusions for Supraglottic Airway Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nalinee Kovitwanawong, Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55-213-08-1-2
Record Dates: First submitted 2014-09-02; First posted 2020-12-11 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Appropriate Affect; Complication of Device Insertion
Keywords: Target Controlled Infusion; Supraglottic airway device; Propofol; Supreme™; ProSeal™; I-gel™; Laryngeal Tube Suction II™
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: 4 second generation of supraglottic airway device
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group SP (Sham Comparator): The Supreme™ group
  Interventions: Drug: Propofol Fresenius
- Group PS (Active Comparator): The ProSeal™ group
  Interventions: Drug: Propofol Fresenius
- Group IG (Active Comparator): The I-gel™ group
  Interventions: Drug: Propofol Fresenius
- Group LT (Active Comparator): The Laryngeal Tube Suction IITM group
  Interventions: Drug: Propofol Fresenius

INTERVENTIONS:
Drug: Propofol Fresenius — final dose of Propofol (mcg/kg) to reach the target effect-site concentration

SUMMARY:
to evaluate and compare the effect-site concentration of propofol with the TCI system for second-generation SGA device insertion between the I-gel™, Supreme™, ProSeal™ and Laryngeal Tube Suction II™.

to determine the hemodynamic changes during insertion of supraglottic devices in patients undergoing elective surgery and any complications after device insertion.

DETAILED DESCRIPTION:
The investigators enrolled ASA physical status I-III patients who were 18-70 years old and scheduled for general anesthesia for elective non-cardiac surgery with SGA devices.Adults with a potentially difficult airway (cervical spine disease, Mallampati classification IV, or a mouth opening less than 2.5 cm.), reactive airway disease, signs of respiratory infection or a plan to remain intubated were excluded from the study. The investigators also excluded patients who had a risk of gastric aspiration or morbid obesity (body mass index > 35 kg/m2).

Patients were randomized into 4 groups (I-gel™, Supreme™, ProSeal™ and Laryngeal Tube Suction II™ SGAs) according to a computer generated randomization list and patients were allocated consecutively. The sample size of each group required 10 patients.

All patients were pre-oxygenated with 100% oxygen. After the administration of 2 µg/ml intravenous fentanyl for 5 minutes, anesthesia was induced with the Schnider pharmacokinetic TCI system. After equilibration of the plasma-site and effect-site concentrations in propofol TCI, 1 of the 4 types of SGA was randomly inserted by two anesthesiologists (resident trainee and staff doctor) who were unaware of the actual plasma concentration of propofol without the use of a muscle relaxant.

The response of each patient determined the effect-site concentration of propofol of the next patient. "No Response" was defined as Laryngeal Mask Airway Insertion Score = 0 and "Response" was defined as Laryngeal Mask Airway Insertion Score ≥ 1. If the insertion of the supraglottic airway device was successful ("No Response"), then the target effect-site concentration was decreased by a step of 0.4 µg/ml. If the insertion failed ("Response"), the target effect-site concentration was increased by the same dose. The patients' responses to LMA insertion was classified by blinded investigators.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III patients.
* Patients 18-70 years old .
* Patients scheduled for general anesthesia for elective non-cardiac surgery with SGA devices.

Exclusion Criteria:

* Adults with a potentially difficult airway (cervical spine disease, Mallampati classification IV, or a mouth opening less than 2.5 cm.).
* Adults with reactive airway disease.
* Adults with signs of respiratory infection or a plan to remain intubated were excluded from the study.
* Excluded patients who had a risk of gastric aspiration or morbid obesity (body mass index > 35 kg/m2).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Tolerability of propofol for supragloqtic airway devices insertion | 2 years
  The effect-site concentration of propofol required to insert supraglottic airway devices.

SECONDARY OUTCOMES:
Blood pressure changes from baseline after insertion of supraglottic devices | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Price of Songkla University, Hat Yai, Changwat Songkhla
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla